CLINICAL TRIAL: NCT07127926
Title: Evaluation of Belumosudil Whole Tablets vs. Crushed Tablets Pharmacokinetics in Patients Suffering From Chronic Graft Versus Host Disease
Brief Title: Evaluation of Belumosudil Whole Tablets vs. Crushed Tablets Pharmacokinetics in Patients Suffering From Chronic GvHD
Status: Not yet recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0041; NCI-2025-05161 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-07-15; First posted 2025-08-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study is to evaluate belumosudil pharmacokinetics of whole tablets and crushed tablets suspended in water in patients suffering from chronic graft-versus-host disease (cGVHD).

DETAILED DESCRIPTION:
Primary Objective:

To evaluate belumosudil pharmacokinetics of whole tablets and crushed tablets suspended in water in patients suffering from chronic graft-versus-host disease (cGVHD).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 years of age with allogeneic HSCT

Exclusion Criteria:

* Receiving an investigational GVHD treatment within 28 days of study entry; (2) active acute GVHD; and (3) taking any medication known to be CYP3A4 inducers.
* Pregnancy is an exclusion criterion for stem cell transplant. Pregnant women are not included in this study. Non-viable neonates will not be included in this study. Patients with cognitive impairments will not be included in this study. Patients aged less than 18 years old will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs | Through study completion; an average of 1 year
  Intra patient change in pharmacokinetic parameters will be determined. In addition, it will be evaluated whether crushing the tablet would have clinically significant change in AUC or Cmax, Tmax, which might impact efficacy or safety of belumosudil based on prior belumosudil pharmacokinetic studies. Due to small number of patients in this study, we don't plan to evaluate the impact of crushed belumosudil tablets pharmacokinetics with long-term outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Amin Alousi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org